CLINICAL TRIAL: NCT07207902
Title: Surveillance or Focal Therapy (SOFT) for Prostate Cancer
Brief Title: Surveillance or Focal Therapy
Acronym: SOFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, David S Finley, MD, Associate Professor of Urology, Kaiser Permanente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB Tracking Number: 057399
Record Dates: First submitted 2025-04-07; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; focal therapy; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men with prostate cancer (Other)
  Interventions: Behavioral: Explainer video

INTERVENTIONS:
Behavioral: Explainer video — 2 minute explainer video on treatment options

SUMMARY:
Patients with newly diagnosed low-intermediate risk prostate cancer often are not advised of all the options in an easy to understand way. This trial will show patients a 2 minute animated Explainer video to better understand their treatment options. Patients will choose their treatment choice (surveillance, focal therapy, or standard treatment option) and we will determine disease related anxiety and decision regret scores.

DETAILED DESCRIPTION:
Low risk prostate cancer is usually monitored with active surveillance (AS). Some evidence suggests no differences in health-related quality of life (HRQoL) and wellness between men undergoing AS and those receiving treatment. However, other studies have shown a significant subset of patients suffers from anxiety or depression related to disease uncertainty. Many patients are given an "all-or-none" binary choice between monitoring or radical treatment. Focal therapy (FT), however, is a potentially less intense treatment option that exists between these extreme choices but is not always presented to the patient due to provider variability. This study seeks to define the proportion of newly diagnosed low/low-int risk prostate cancer patients who elect to pursue HIFU or surveillance when presented with all treatment options devoid of persuasive rhetoric using an animated explainer video. Secondary outcomes will include anxiety score and decision regret.

ELIGIBILITY:
Inclusion Criteria:

* Gleason 3+3 (GG 1) or 3+4 (GG2)
* ≤4 cores
* T1c-T2
* Prostate < 60cc
* MRI non-focal or PIRADS 3-4 in peripheral gland
* Absence of significant anterior disease

Exclusion Criteria:

* Anal stenosis
* Prostatic calfcifations
* Latex allergy
* Gleason grade group 3-5
* Multifocal or anterior disease
* Prostate > 60 cc

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men with prostate cancer
Enrollment: 400 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment choice | 12 months
  Incidence of surveillance, focal therapy, or other treatment choice

SECONDARY OUTCOMES:
Decision regret and anxiety scale | 12 months
  Anxiety and Decision Regret Score

CONTACTS AND LOCATIONS:
Overall Officials: David S Finley, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided